CLINICAL TRIAL: NCT05552911
Title: Clinical Prognosis and Influencing Factors of Drug-coated Balloon Therapy in Patients With Coronary In-stent Restenosis and de Novo Coronary Lesions
Brief Title: Drug-coated Balloon Therapy for In-stent Restenosis and de Novo Coronary Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, Department of cardiovascular, Director of CCU, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 19
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Coronary Heart Disease
Keywords: Drug-coated balloon; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- De novo coronary lesions: cutting balloon group: De novo coronary lesions were pretreated with a cutting balloon and then treated with a drug-coated balloon.
  Interventions: Procedure: Pretreatment strategies before drug balloon therapy
- De novo coronary lesions: non-cutting balloon group: De novo coronary lesions were pretreated with a non-cutting (Compliance balloon or/and non-compliant balloon) balloon and then treated with a drug-coated balloon.
  Interventions: Procedure: Pretreatment strategies before drug balloon therapy
- In-stent restenosis: Type-I: Body stenosis: restenosis of the stent body, not beyond the edge of the stent.The lesions were pretreated with balloon dilation and then treated with drug-coated balloons.
  Interventions: Procedure: Different types of in-stent restenosis were treated with drug-coated balloons
- In-stent restenosis: Type-II: Marginal stenosis type: restenosis at the edge of the stent, stenosis ≥50% within 5mm of the stent edge, which can continue into the stent.The lesions were pretreated with balloon dilation and then treated with drug-coated balloons.
  Interventions: Procedure: Different types of in-stent restenosis were treated with drug-coated balloons
- In-stent restenosis:Type-III: Diffuse proliferative type: the lesion extends to the whole scaffold body and beyond the edge of both ends.The lesions were pretreated with balloon dilation and then treated with drug-coated balloons.
  Interventions: Procedure: Different types of in-stent restenosis were treated with drug-coated balloons
- In-stent restenosis:Type-IV: Complete occlusion type: complete occlusion in the stent.The lesions were pretreated with balloon dilation and then treated with drug-coated balloons.
  Interventions: Procedure: Different types of in-stent restenosis were treated with drug-coated balloons

INTERVENTIONS:
Procedure: Pretreatment strategies before drug balloon therapy — Preconditioning strategies for the treatment of in de novo coronary lesions using drug-coated balloons.
  Groups: De novo coronary lesions: cutting balloon group; De novo coronary lesions: non-cutting balloon group
Procedure: Different types of in-stent restenosis were treated with drug-coated balloons — A new classification method of ISR lesions was proposed to observe the clinical prognosis of different ISR lesions treated with drug-coated balloon.
  Groups: In-stent restenosis: Type-I; In-stent restenosis: Type-II; In-stent restenosis:Type-III; In-stent restenosis:Type-IV

SUMMARY:
This was a single-center, prospective, open-label, observational study. Patients with coronary artery disease confirmed by coronary angiography and treated with drug-coated balloon catheter alone for target vessels were enrolled in the Cardiology Department of our hospital in January 2022. The primary endpoint was late lumen loss within 12±3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years with coronary heart disease;
2. If the target lesion stenosis ≥70% is complicated with angina pectoris or evidence of myocardial ischemia, DCB should be administered;
3. Residual lumen diameter stenosis ≤30% after lesion pretreatment and DCB, no vessel dissection, or type A or B dissection, and TIMI blood flow level 3;
4. Target lesions were treated with DCB for the first time.

Exclusion Criteria:

1. Intraoperative implantation of salvage stent in DCB;
2. Acute myocardial infarction occurred within 1 week after DCB operation;
3. Less than 3 months of dual antiplatelet therapy after DCB operation, or more than 1 month of discontinuation of antiplatelet therapy;
4. The position of the stent could not be determined by coronary angiography.
5. Desmovascular disease or left main artery disease;
6. Atrial fibrillation;
7. Patients with severe heart failure, valvular heart disease, renal insufficiency, severe infection and autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with coronary heart disease by coronary angiography and treated with DCB alone in the Department of Cardiology of our hospital since January 2022 were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
LLL of 12±3 months after surgery | 12±3 months after surgery
  Late lumen loss of 12±3 months after surgery

SECONDARY OUTCOMES:
MACE event 12 months after surgery | 12 months after surgery
  The incidence of MACE events (target vessel revascularization, target vessel myocardial infarction, cardiac death) at 12 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No